CLINICAL TRIAL: NCT04961502
Title: Humoral and Cellular Responses to Vaccination Against Coronavirus Disease 2019 (COVID-19) in the Very Elderly Living in Geriatric Institutions
Acronym: COGEVAX-BIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2021-A00051-40
Record Dates: First submitted 2021-06-04; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Elderly People Institutionalized in Long-term Care Services
Keywords: mRNA BNT162b2 vaccine; Coronavirus desease 2019 (Covid-19); anti-RBD IgG; vaccine antibodies; blood sample
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 3 blood samples taken to compare the immunization response of the elderly with that of younger adults (priority caregivers)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderly person (Experimental): Three blood sample: the first carried out before the anti-COVID-19 vaccination; the second shortly before the vaccination booster injection and the third approximately two months after the first vaccine injection
  Interventions: Biological: Blood test to describe the humoral and cellular response to vaccination BNT162b2 in the elderly
- Younger adults (priority caregivers) (Active Comparator): Three blood sample: the first carried out before the anti-COVID-19 vaccination; the second shortly before the vaccination booster injection and the third approximately two months after the first vaccine injection
  Interventions: Biological: Blood test to describe the humoral and cellular response to vaccination BNT162b2 in the elderly

INTERVENTIONS:
Biological: Blood test to describe the humoral and cellular response to vaccination BNT162b2 in the elderly — 3 blood samples taken to compare the immunization response of the elderly with that of younger adults (priority caregivers): the first carried out before the anti-Coronavirus Disease 2019 (COVID-19) vaccination; the second shortly before the vaccination booster injection and the third approximately two months after the first vaccine injection

SUMMARY:
The main objective of this study is to describe the humoral and cellular response to BNT162b2 vaccination in people over age 75 institutionalized in the long-term care units of the Paris Public Hospitals (APHP)

DETAILED DESCRIPTION:
This is an interventional study with minimal risk and constraints, multicenter with biological collection. Two populations are studied: patients and members of care staff.

The following data will be collected:

* For patients and staff: age, gender, existence of Coronavirus Disease 2019 (COVID-19) infection and whether or not it is symptomatic and date of first positive RT-PCR test, medical history
* For patients: nutritional status (loss of appetite, weight loss, body mass index, albuminemia)

Vaccination antibodies are measured using 3 blood sample:

The first carried out before the anti-Coronavirus Disease 2019 (COVID-19) vaccination; the second on D21 (shortly before the vaccination booster injection) and the third on D50-54.

In addition, during the first sample, assays will be carried out informing us of your nutritional and inflammatory status.

ELIGIBILITY:
Inclusion Criteria for patients:

* Person aged 75 and over,
* Hospitalized in a long-term care unit participating in the study,
* Having agreed to be vaccinated with the BNT162b2 vaccine as part of the phase 1 vaccination campaign defined by the health authorities,
* Not having received any other vaccination or corticosteroid treatment during the 3 weeks preceding the start of the study,
* Having given their written consent to participate in the study, or having not expressed their opposition to participating and whose legal guardian has given their consent.

Inclusion Criteria for younger adults (priority care staff):

* Staff who have agreed to be vaccinated with the BNT162b2 vaccine as part of the phase 1 vaccination campaign defined by the health authorities,
* Not having received any other vaccination or corticosteroid treatment during the 3 weeks preceding the start of the study,
* Having given their written consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Measure plasma concentration of anti-RBD IgG antibodies in elderly using SARS-CoV-2 IgG II Quant assay technique (Abbott) | 50 days

SECONDARY OUTCOMES:
Measure plasma concentration of anti-RBD IgG antibodies in younger adults using SARS-CoV-2 IgG II Quant assay technique (Abbott) | 50 days
Assess the percentage of patients with previous COVID-19 infection prior to vaccination | At inclusion

OTHER OUTCOMES:
Assessment the percentage of patients who developed anti-RBD antibodies after vaccination by blood sample | 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Joël Belmin, MD PhD, Study Chair — Geriatric Department, Charles Foix hospital
Locations (1):
- Geriatric Department, Charles Foix hospital, Ivry-sur-Seine, IIe-de-France, France